CLINICAL TRIAL: NCT02439112
Title: Early Initiated Individualized Physical Training in Newly Diagnosed Multiple Myeloma Patients; Effects on Physical Function, Physical Activity, Quality of Life, Pain, and Bone Disease.
Brief Title: Exercise in Patients With Multiple Myeloma
Acronym: EMMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Odense University Hospital (Other); Region Zealand (Other); Region of Southern Denmark (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Reum,fys/ergo 1
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Multiple Myeloma
Keywords: Exercise; Physical Function; Physical Activity; Quality of Life; Pain; Bone Disease
MeSH Terms: conditions — Multiple Myeloma; Motor Activity; Pain; Bone Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Active Comparator): Supervised exercise combined with home based exercise and physical activity
  Interventions: Other: Exercise
- Control (No Intervention): Usual care consisting of advice regarding exercise, physical activity, person lifting and moving.

INTERVENTIONS:
Other: Exercise — 8 supervised in-hospital training sessions in a period of 10 weeks. On a general level, the intervention will follow the Danish physical activity guidelines for elderly >65 years (Sundhedsstyrelsen 2011, see link) and consist of strength exercise, aerobic exercise and physical activity.
  Bone involvement will taken into consideration in all parts of the exercise program by excluding and including specific exercises and mode of exercise according to location and extent of bone involvement (Galvão 2011; Cormie 2013)
  Arms: Exercise

SUMMARY:
The overall aim is to examine whether early initiated, individualized exercise training in patients newly diagnosed with multiple myeloma, irrespective of age and current performance status, will be beneficial for the patients´physical function, level of physical activity and quality of life, pain and bone disease.

The investigators will examine the effect of supervised in-hospital exercise training sessions combined with home-based exercise training, initiated at time of diagnosis. The outcomes of interest are physical function, level of physical activity, QOL, pain and bone disease.

Furthermore, to describe the disease in patients with newly diagnosed MM in relation to physical function, level of physical activity, QOL, pain and bone condition at time of diagnosis.

The investigators hypotheses are:

* Individualized exercise starting at time of diagnosis will have positive effects on physical function, physical activity, QOL and pain.
* Individualized exercise starting at time of diagnosis will have positive effects on bone disease (bone markers), bone mineral density (BMD) and lean body mass.
* A higher level of physical function is associated with a higher level of physical activity, less pain, better QOL, and higher BMD and lean body mass.

DETAILED DESCRIPTION:
Background Physical exercise for haematological patients is a relevant complementary treatment, including in patients with multiple myeloma (MM) (Jones 2013). In hematological cancer, exercise is feasible, safe and beneficial in numerous aspects (aerobic capacity, muscle strength, quality of life (QOL), fatigue, psychosocial wellbeing, treatment-related symptoms and body composition, before, during and after stem cell transplantation (Persoon 2013; Haren 2013). Still the evidence for the value of exercise in hematological diseases is sparse, in general and to specific diagnoses (Jones 2013; Fong 2014; Liu 2009). Patients with MM may differ from other hematological diseases, by poorer functional status due to skeletal related pain, affected QOL and immune function, but also in return to work and in risk of disability pension, and furthermore physical performance and the time of being physical active is diminished throughout the treatment course and patients do not meet physical activity guidelines (Coleman 2004; Jones 2004; Craike 2013). Hence, there is a need to examine the effect of exercise to be able to give evidence based recommendations on exercise in MM patients.

In Denmark, 320 patients are diagnosed with MM annually. The median age at diagnosis is 68-71 years, and the incidence is increasing with age. The prevalence increases due to the aging population and improved survival because of improvement in medical treatment (Kyle 2007; Sihori 2006 & 2004; Alexander 2007; Kumar 2008 & 2014). Typically, the patient presents with bone pain, anaemia, renal failure, recurrent infections, or for some patients it is detected by chance through screening of blood or urine. Bone pain is caused by osteolytic destructions which also may lead to pathological fractures.

When diagnosed, most patients (80%) will have symptomatic disease and will need start treatment. The medical treatment for MM has two aims. Firstly, anti-myeloma systemic therapy aims at reducing tumor burden and to prolong disease free survival, and overall survival, and secondly, supportive care aims at preventing serious morbidity from disease complications. Younger patients (<65-70 year) are treated with high dose chemotherapy with stem cell support (HDT). Elderly patients receive less intensive, yet still effective treatments that include novel agents (bortezomib, thalidomide). Painful bone lytic lesions may be treated with radiation therapy. Patients receive i.v. bisphosphonates to reduce the risk of progressive bone disease and fractures (Rosen 2003; Morgan 2011).

Patients with MM (receiving HDT) perceive different symptoms (sleep and mood disturbances, diminished functional performance, pain, shortness of breath, distress, sadness and difficulty paying attention. Symptoms are interrelated and a vicious circle may be present (Coleman 2011; Anderson 2007).

Literature review: Exercise in patients with MM Only 3 RCT studies (Coleman 2003 & 2008 & 2012) and 1 single arm pilot study (Groeneveldt 2013) regarding the effect of exercise in patients with MM have been identified. Coleman investigated patients undergoing tandem autologous peripheral blood stem cell transplantation with no risk of fracture, while Groeneveldt investigated MM survivors. All the exercise programs were individualized and home-based, although one study also included weekly supervised training the first three months and monthly the following 3 months. The exercise programs, all compromising stretching, aerobic training and strength resistance training, had a duration of 6 months, and 3 of them started during induction and HDT. The controls were advised to walk 20 minutes 3 times a week.

The single arm pilot study in MM survivors showed significant positive changes in QOL, fatigue and muscle strength, but not in aerobic fitness. Positive, although not significant, changes were seen regarding anxiety/depression. In the studies of Coleman et al. there was a trend towards less decline in aerobic capacity/physical performance in the exercise group compared to the control group. Lean body weight (per month) were significantly increased among those exercising compared to controls. Over the 6 months period strength and lean body weight increased and they perceived less fatigue, better mood and more night time sleep than the controls. Trends of physiologic benefits regarding stem cell collection and transfusions during transplantation were shown.

One Coleman study showed statistical significant changes during the treatment course; decline in physical performance, increase in perceived fatigue, and negative effect on the night sleep, both in the exercise group or the control group. There was no statistical or clinical significant differences in any of the investigated outcomes between the exercise group and the control group at all test times prior to chemotherapy, 10-12 weeks later and 15-16 weeks after stem cell collection. The lack of significant results can be due to poor compliance (based on self-reported activity summary with no results reported in the paper), no structured supervision throughout the exercise intervention and perhaps inadequate intensity in relation to an effect in aerobic capacity. Moreover, the Arkansas anti-myeloma Total Therapy Program is a highly intensive chemotherapy that is not comparable with the induction regimens that are used in Denmark. This highly intensive treatment may very well counteract the benefits of physical training. However, it is noteworthy, that the exercise group had a better physical performance than the control group, although not significant. Importantly, the exercise programs were feasible, acceptable and safe. The performed studies have different shortcomings, such as small study populations, lack of control group, lack of supervised training, no description of whether the assessor was blinded, and inadequate description of the intervention.

In summary, exercise is found to be safe and feasible in patients with MM during induction and HDT, and after discharge. There is a gap in the literature concerning elderly patients with MM and in general in patients treated with less intensive regimens than HDT.

The effect of exercise on physical function needs further examination, especially because the broad group of patients with MM also compromises elderly patients, making exercise even more relevant as a complementary treatment early in the disease course in order to maintain physical function. Because of the nature of the disease involving the bones, it is believed that exercise may be beneficial for maintaining MM patients´ both regarding physical function and bone loss, as in the older population (Chin 2008) and in patients with osteoporosis (Hagen 2011; Howe 2011) or as found in the encouraging results regarding bone health among cancer survivors (Winters-Stone 2010). The literature suggests that combined training is beneficial in order to maintain or increase BMD and lean body mass among patients with prostate cancer or breast cancer (Bolam 2012; Cormie 2014), among post menopausal women (Martyn-St James 2008 & 2009; Palombaro 2006) and among elderly (Gómez-Cabello 2012). Change in bone markers as an effect of exercise have also been investigated, although in different exercise protocols. The results from healthy women and men are promising. Bone formation markers are significantly increased, without significant changes in bone resorption markers (Shibata 2003; Karabulut 2011). OQL, in a disease specific perspective, needs attention since exercise can improve QOL (Persoon 2013; Haren 2013; Mishra 2012 & 2012), and since bone pain is a major problem in patients with MM, it is relevant to investigate pain as a separate outcome. It has been demonstrated, that breast cancer survivors meeting physical activity guidelines are significant less likely to report above-average pain than breast cancer survivors not meeting physical activity guidelines, and those who always have been physically active report less pain than inactive women (Forsythe 2013). Griffith (2009) have found, that cancer patients report a lower pain level, if they become more physically active (adjusted for age, cancer diagnosis, pretest pain, pretest physical activity/physical functioning), but Forsythe (2013) have demonstrated unchanged pain level despite increase in physical activity. These results make it even more important to investigate pain in the investigators set up. Physical functioning will have impact on the level of physical activity, which has importance in a long term perspective, but to the investigators knowledge the level of physical activity has not been investigated in patients with MM neither in a prospective design nor with objective measurements.

Recruitment All patients with newly diagnosed MM at Roskilde Hospital and Odense University Hospital will be screened for eligibility on the basis of inclusion and exclusion criteria, at their first appointment with the physician (hematologist) at time of diagnosis.

If eligible, the physician will both briefly inform the patient about the project, and give the written participation information. Before the next consultation (typically after 2-3 days), the investigator will call the patient with further information and address any questions the patient may have regarding the project before written informed consent is obtained.If not eligible or the patient does not want to participate, the patient will be registered only by the reason for exclusion.

Design After inclusion the patients will be randomized 1:1 into an intervention group or control group. The participants will be block randomized and stratified to treatment (planned HDT versus (vs.) non-intensive treatment), performance status (PFS 0-1 vs. PFS≥2) (Oken 1982), and study site (Roskilde vs. Odense). The intervention will start at day 8 (in the 2nd week) after start of treatment unless safety reasons make it necessary to postpone start of exercise. The measurements at all time points will be conducted by experienced, educated investigators (physiotherapists). Measurements will preferably be conducted by the same physiotherapist at each site.

Power calculation The number of patients to be included has been determined by a power calculation, with a significance level, α = 0.05 and 80% power, β = 0.20 and a minimum clinical difference of mean(SD) 7 kg(13.1) in the knee extensor strength (Groeneveldt 2013), which is the primary outcome (corresponding to an increase of approximately 23 %). The number of patients needed, can be estimated to 44 patients in each group (intervention and control).

Statistical analysis It will be tested whether data follow a normal distribution.The following description is based on the assumption that data is normally distributed. For continuous data in an interval scale, mean(sd) will be used and for data in an ordinal scale, median(range) and quartiles will be used to describe data. Differences within group between test times and between groups at all test times will be examined by t-test. The significance level is set to p<0,05. The analysis will be conducted in accordance with ITT.

To test the investigators hypothesis on the primary outcome (knee extensor strength), t-test will be used and the standard error of the mean difference will be calculated. A mean difference of 7 kg is considered clinical significant, and if this is obtained H0 can be rejected.

To investigate associations between physical function and physical activity, QOL, pain, lean body mass, BMD, and bone markers, scatter plots will be used. If linear correlations exist, the correlations coefficients will be calculated. The correlation will be tested with Fisher´s z transformation and 95%CI will be formed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Multiple Myeloma requiring treatment.
* The patient must be able to speak and understand Danish and be able to give his/her informed consent.

Exclusion Criteria:

* Patients with spinal cord compression
* Unstable vertebral fracture (SINS score >12) (52)
* Untreated cardiac failure and untreated cardiac arrythmia
* Severe chronic cardiac failure (NYHA 3-4)
* Other severe comorbidity that will not allow physical training, e.g. neurological or uncompensated liver failure and psychological or psychiatric disorder that will not allow compliance in physical training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2020-02-05 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in isometric knee extension strength measured by handhold dynamometer | From baseline to follow-up after 11 weeks
  kilogram and newton

SECONDARY OUTCOMES:
Change in isometric knee extension strength measured by handhold dynamometer | Baseline and follow-up after 6 months and 12 months
  kilogram and newton
Change in lower limb strength measured by Sit-to-Stand Test | Baseline and follow-up after 11 weeks, 6 months and 12 months
  Functional test of lower limb strength
Change in grip strength measured by hand dynamometer | Baseline and follow-up after 11 weeks, 6 months and 12 months
  kilogram
Change in aerobic capacity measured by 6 Minutes Walk Test | Baseline and follow-up after 11 weeks, 6 months and 12 months
  Test of submaximal aerobic capacity
Change in Quality of Life assessed by self-reported questionnaire | Baseline and follow-up after 11 weeks, 6 months and 12 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC QLQ-C30) and The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20) (68)
Change in pain assessed by self-reported questionnaire | Baseline and follow-up after 11 weeks, 6 months and 12 months
  Brief Pain Inventory (BPI) (70,71)
Change in level of physical activity measured by accelerometer | Baseline and follow-up after, 4 weeks, 7 weeks, 11 weeks, 6 months and 12 months
  Measured objectively by accelerometer (ActivPal) in periods of 5 days
Change in bone disease - dynamic markers | Baseline and follow-up after 11 weeks, 6 months and 12 months
  Osteoblast and osteoclast activity measured by dynamic markers (PINP and CTX-1) of bone metabolism in serum.
Change in bone disease - Bone Mineral Density assessed by DEXA scans | Baseline and follow-up after 6 months and 12 months
  Dual-Energy X-ray Absorptiometry (DEXA)
Change in Lean Body Mass assessed by DEXA scans | Baseline and follow-up after 11 weeks, 6 months and 12 months
  Dual-Energy X-ray Absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Rikke F Larsen, Ph.d., Principal Investigator — Department of Hematology, Odense University Hospital, DK; Niels Abildgaard, Professor, Study Chair — Department of Hematology, Odense University Hospital, DK and University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones LW, Alfano CM. Exercise-oncology research: past, present, and future. Acta Oncol. 2013 Feb;52(2):195-215. doi: 10.3109/0284186X.2012.742564. Epub 2012 Dec 17. PMID 23244677
- [Background] Persoon S, Kersten MJ, van der Weiden K, Buffart LM, Nollet F, Brug J, Chinapaw MJ. Effects of exercise in patients treated with stem cell transplantation for a hematologic malignancy: a systematic review and meta-analysis. Cancer Treat Rev. 2013 Oct;39(6):682-90. doi: 10.1016/j.ctrv.2013.01.001. Epub 2013 Feb 26. PMID 23485478
- [Background] van Haren IE, Timmerman H, Potting CM, Blijlevens NM, Staal JB, Nijhuis-van der Sanden MW. Physical exercise for patients undergoing hematopoietic stem cell transplantation: systematic review and meta-analyses of randomized controlled trials. Phys Ther. 2013 Apr;93(4):514-28. doi: 10.2522/ptj.20120181. Epub 2012 Dec 6. PMID 23224217
- [Background] Fong DY, Ho JW, Hui BP, Lee AM, Macfarlane DJ, Leung SS, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Physical activity for cancer survivors: meta-analysis of randomised controlled trials. BMJ. 2012 Jan 30;344:e70. doi: 10.1136/bmj.e70. PMID 22294757
- [Background] Liu RD, Chinapaw MJ, Huijgens PC, van Mechelen W. Physical exercise interventions in haematological cancer patients, feasible to conduct but effectiveness to be established: a systematic literature review. Cancer Treat Rev. 2009 Apr;35(2):185-92. doi: 10.1016/j.ctrv.2008.09.008. Epub 2008 Nov 11. PMID 19004560
- [Background] Coleman EA, Goodwin JA, Kennedy R, Coon SK, Richards K, Enderlin C, Stewart CB, McNatt P, Lockhart K, Anaissie EJ. Effects of exercise on fatigue, sleep, and performance: a randomized trial. Oncol Nurs Forum. 2012 Sep;39(5):468-77. doi: 10.1188/12.ONF.468-477. PMID 22940511
- [Background] Jones LW, Courneya KS, Vallance JK, Ladha AB, Mant MJ, Belch AR, Stewart DA, Reiman T. Association between exercise and quality of life in multiple myeloma cancer survivors. Support Care Cancer. 2004 Nov;12(11):780-8. doi: 10.1007/s00520-004-0668-4. PMID 15322968
- [Background] Craike M, Hose K, Livingston PM. Physical activity participation and barriers for people with multiple myeloma. Support Care Cancer. 2013 Apr;21(4):927-34. doi: 10.1007/s00520-012-1607-4. Epub 2012 Oct 2. PMID 23052913
- [Background] Kyle RA, Rajkumar SV. Epidemiology of the plasma-cell disorders. Best Pract Res Clin Haematol. 2007 Dec;20(4):637-64. doi: 10.1016/j.beha.2007.08.001. PMID 18070711
- [Background] Sirohi B, Powles R. Epidemiology and outcomes research for MGUS, myeloma and amyloidosis. Eur J Cancer. 2006 Jul;42(11):1671-83. doi: 10.1016/j.ejca.2006.01.065. Epub 2006 Jul 25. PMID 16870424
- [Background] Alexander DD, Mink PJ, Adami HO, Cole P, Mandel JS, Oken MM, Trichopoulos D. Multiple myeloma: a review of the epidemiologic literature. Int J Cancer. 2007;120 Suppl 12:40-61. doi: 10.1002/ijc.22718. PMID 17405120
- [Background] Sirohi B, Powles R. Multiple myeloma. Lancet. 2004 Mar 13;363(9412):875-87. doi: 10.1016/S0140-6736(04)15736-X. PMID 15031034
- [Background] Kumar SK, Dispenzieri A, Lacy MQ, Gertz MA, Buadi FK, Pandey S, Kapoor P, Dingli D, Hayman SR, Leung N, Lust J, McCurdy A, Russell SJ, Zeldenrust SR, Kyle RA, Rajkumar SV. Continued improvement in survival in multiple myeloma: changes in early mortality and outcomes in older patients. Leukemia. 2014 May;28(5):1122-8. doi: 10.1038/leu.2013.313. Epub 2013 Oct 25. PMID 24157580
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Morgan GJ, Child JA, Gregory WM, Szubert AJ, Cocks K, Bell SE, Navarro-Coy N, Drayson MT, Owen RG, Feyler S, Ashcroft AJ, Ross FM, Byrne J, Roddie H, Rudin C, Cook G, Jackson GH, Wu P, Davies FE; National Cancer Research Institute Haematological Oncology Clinical Studies Group. Effects of zoledronic acid versus clodronic acid on skeletal morbidity in patients with newly diagnosed multiple myeloma (MRC Myeloma IX): secondary outcomes from a randomised controlled trial. Lancet Oncol. 2011 Aug;12(8):743-52. doi: 10.1016/S1470-2045(11)70157-7. Epub 2011 Jul 21. PMID 21771568
- [Background] Rosen LS, Gordon D, Kaminski M, Howell A, Belch A, Mackey J, Apffelstaedt J, Hussein MA, Coleman RE, Reitsma DJ, Chen BL, Seaman JJ. Long-term efficacy and safety of zoledronic acid compared with pamidronate disodium in the treatment of skeletal complications in patients with advanced multiple myeloma or breast carcinoma: a randomized, double-blind, multicenter, comparative trial. Cancer. 2003 Oct 15;98(8):1735-44. doi: 10.1002/cncr.11701. PMID 14534891
- [Background] Coleman EA, Goodwin JA, Coon SK, Richards K, Enderlin C, Kennedy R, Stewart CB, McNatt P, Lockhart K, Anaissie EJ, Barlogie B. Fatigue, sleep, pain, mood, and performance status in patients with multiple myeloma. Cancer Nurs. 2011 May-Jun;34(3):219-27. doi: 10.1097/NCC.0b013e3181f9904d. PMID 21522061
- [Background] Coleman EA, Coon S, Hall-Barrow J, Richards K, Gaylor D, Stewart B. Feasibility of exercise during treatment for multiple myeloma. Cancer Nurs. 2003 Oct;26(5):410-9. doi: 10.1097/00002820-200310000-00012. PMID 14710804
- [Background] Coleman EA, Coon SK, Kennedy RL, Lockhart KD, Stewart CB, Anaissie EJ, Barlogie B. Effects of exercise in combination with epoetin alfa during high-dose chemotherapy and autologous peripheral blood stem cell transplantation for multiple myeloma. Oncol Nurs Forum. 2008 May;35(3):E53-61. doi: 10.1188/08.ONF.E53-E61. PMID 18467280
- [Background] Groeneveldt L, Mein G, Garrod R, Jewell AP, Van Someren K, Stephens R, D'Sa SP, Yong KL. A mixed exercise training programme is feasible and safe and may improve quality of life and muscle strength in multiple myeloma survivors. BMC Cancer. 2013 Jan 24;13:31. doi: 10.1186/1471-2407-13-31. PMID 23347597
- [Background] Chin A Paw MJ, van Uffelen JG, Riphagen I, van Mechelen W. The functional effects of physical exercise training in frail older people : a systematic review. Sports Med. 2008;38(9):781-93. doi: 10.2165/00007256-200838090-00006. PMID 18712944
- [Background] Hagen KB, Dagfinrud H, Moe RH, Osteras N, Kjeken I, Grotle M, Smedslund G. Exercise therapy for bone and muscle health: an overview of systematic reviews. BMC Med. 2012 Dec 19;10:167. doi: 10.1186/1741-7015-10-167. PMID 23253613
- [Background] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Background] Winters-Stone KM, Schwartz A, Nail LM. A review of exercise interventions to improve bone health in adult cancer survivors. J Cancer Surviv. 2010 Sep;4(3):187-201. doi: 10.1007/s11764-010-0122-1. Epub 2010 Apr 7. PMID 20373041
- [Background] Bolam KA, Galvao DA, Spry N, Newton RU, Taaffe DR. AST-induced bone loss in men with prostate cancer: exercise as a potential countermeasure. Prostate Cancer Prostatic Dis. 2012 Dec;15(4):329-38. doi: 10.1038/pcan.2012.22. Epub 2012 Jun 26. PMID 22733158
- [Background] Cormie P, Galvao DA, Spry N, Joseph D, Taaffe DR, Newton RU. Functional benefits are sustained after a program of supervised resistance exercise in cancer patients with bone metastases: longitudinal results of a pilot study. Support Care Cancer. 2014 Jun;22(6):1537-48. doi: 10.1007/s00520-013-2103-1. Epub 2014 Jan 15. PMID 24424484
- [Background] Martyn-St James M, Carroll S. A meta-analysis of impact exercise on postmenopausal bone loss: the case for mixed loading exercise programmes. Br J Sports Med. 2009 Dec;43(12):898-908. doi: 10.1136/bjsm.2008.052704. Epub 2008 Nov 3. PMID 18981037
- [Background] Martyn-St James M, Carroll S. Meta-analysis of walking for preservation of bone mineral density in postmenopausal women. Bone. 2008 Sep;43(3):521-31. doi: 10.1016/j.bone.2008.05.012. Epub 2008 May 26. PMID 18602880
- [Background] Palombaro KM. Effects of walking-only interventions on bone mineral density at various skeletal sites: a meta-analysis. J Geriatr Phys Ther. 2005;28(3):102-7. doi: 10.1519/00139143-200512000-00006. PMID 16386172
- [Background] Gomez-Cabello A, Ara I, Gonzalez-Aguero A, Casajus JA, Vicente-Rodriguez G. Effects of training on bone mass in older adults: a systematic review. Sports Med. 2012 Apr 1;42(4):301-25. doi: 10.2165/11597670-000000000-00000. PMID 22376192
- [Background] Shibata Y, Ohsawa I, Watanabe T, Miura T, Sato Y. Effects of physical training on bone mineral density and bone metabolism. J Physiol Anthropol Appl Human Sci. 2003 Jul;22(4):203-8. doi: 10.2114/jpa.22.203. PMID 12939536
- [Background] Karabulut M, Bemben DA, Sherk VD, Anderson MA, Abe T, Bemben MG. Effects of high-intensity resistance training and low-intensity resistance training with vascular restriction on bone markers in older men. Eur J Appl Physiol. 2011 Aug;111(8):1659-67. doi: 10.1007/s00421-010-1796-9. Epub 2011 Jan 5. PMID 21207053
- [Background] Mishra SI, Scherer RW, Snyder C, Geigle PM, Berlanstein DR, Topaloglu O. Exercise interventions on health-related quality of life for people with cancer during active treatment. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD008465. doi: 10.1002/14651858.CD008465.pub2. PMID 22895974
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Forsythe LP, Alfano CM, George SM, McTiernan A, Baumgartner KB, Bernstein L, Ballard-Barbash R. Pain in long-term breast cancer survivors: the role of body mass index, physical activity, and sedentary behavior. Breast Cancer Res Treat. 2013 Jan;137(2):617-30. doi: 10.1007/s10549-012-2335-7. Epub 2012 Dec 15. PMID 23242613
- [Background] Griffith K, Wenzel J, Shang J, Thompson C, Stewart K, Mock V. Impact of a walking intervention on cardiorespiratory fitness, self-reported physical function, and pain in patients undergoing treatment for solid tumors. Cancer. 2009 Oct 15;115(20):4874-84. doi: 10.1002/cncr.24551. PMID 19637345
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Anderson KO, Giralt SA, Mendoza TR, Brown JO, Neumann JL, Mobley GM, Wang XS, Cleeland CS. Symptom burden in patients undergoing autologous stem-cell transplantation. Bone Marrow Transplant. 2007 Jun;39(12):759-66. doi: 10.1038/sj.bmt.1705664. Epub 2007 Apr 16. PMID 17438588
- [Background] Galvao DA, Taaffe DR, Cormie P, Spry N, Chambers SK, Peddle-McIntyre C, Baker M, Denham J, Joseph D, Groom G, Newton RU. Efficacy and safety of a modular multi-modal exercise program in prostate cancer patients with bone metastases: a randomized controlled trial. BMC Cancer. 2011 Dec 13;11:517. doi: 10.1186/1471-2407-11-517. PMID 22166044
- [Background] Cormie P, Newton RU, Spry N, Joseph D, Taaffe DR, Galvao DA. Safety and efficacy of resistance exercise in prostate cancer patients with bone metastases. Prostate Cancer Prostatic Dis. 2013 Dec;16(4):328-35. doi: 10.1038/pcan.2013.22. Epub 2013 Aug 6. PMID 23917308
- [Derived] Larsen RF, Jarden M, Minet LR, Frolund UC, Moller S, Abildgaard N. Physical function in patients newly diagnosed with multiple myeloma; a Danish cohort study. BMC Cancer. 2020 Mar 3;20(1):169. doi: 10.1186/s12885-020-6637-6. PMID 32126972
- [Derived] Larsen RF, Jarden M, Minet LR, Frolund UC, Abildgaard N. Supervised and home-based physical exercise in patients newly diagnosed with multiple myeloma-a randomized controlled feasibility study. Pilot Feasibility Stud. 2019 Nov 12;5:130. doi: 10.1186/s40814-019-0518-2. eCollection 2019. PMID 31741745